CLINICAL TRIAL: NCT01560585
Title: Open Label Study of Isotretinoin in Mild to Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Adverse events in 2/3 participants; study was halted but not restarted after this due to insufficnet funds as well
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Alan Lerner, MD, Director, Brain Health and Memory Center, Neurological Institute, University Hospitals Cleveland Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISOTRT-01
Record Dates: First submitted 2012-03-15; First posted 2012-03-22 (Estimated); Results first posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-05

CONDITIONS: Alzheimer's Disease
Keywords: Isotretinoin; Alzheimer's disease; Dementia; Retinoid
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Isotretinoin

STUDY DESIGN:
Masking Description: "open label study" before being prematurely terminated
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open label (Experimental): All participants will receive Isotretinoin for 24 weeks
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Isotretinoin — Isotretinoin 0.5 mg per kilogram body weight (rounded to nearest 10 mg) per day for 24 weeks

SUMMARY:
This is an open label study of isotretinoin, a medication which is FDA approved for treatment of other conditions to determine initial safety in Alzheimer's disease.

DETAILED DESCRIPTION:
Retinoids have some relevant characteristics that could be considered useful in treating AlZheimer's disease. These include anti-inflammatory properties, possible anti-amyloid formation proeprties and inhibition of cell cycle properties

ELIGIBILITY:
Inclusion Criteria:

* Probable AD by DSM IV and NINCDS-ADRDA criteria
* Females must be surgically sterile (bilateral tubal ligation, both ovaries removed or hysterectomy) or post-menopausal for at least 2 years.
* > 50 years of age
* Residing in the community at baseline (includes assisted living facilities, long-term care nursing facilities)
* Mini Mental State Examination at screen of 12-26 (inclusive)
* No medical contraindications to study participation
* Fluent in English at least 8 years of education.
* Supervision available for study medication. Caregiver/study partner to accompany participant to all visits. Study partner must have direct contact with the participant > 2 days/week
* Able to ingest oral medication.
* Neuroimaging (CT or MRI or PET) consistent with the diagnosis of AD at some time after the onset of the memory decline.
* Clinical laboratory values must be within normal limits or, if abnormal, must be judged to be clinically insignificant by the investigator
* Stable use of cholinesterase inhibitors and memantine is permitted if doses are stable for 3 months prior to enrollment. Dose should be stable throughout the study unless it is clinically necessary to adjust the medication.
* Stable use of anti-depressants is permitted if doses are stable for 3 months prior to enrollment. Dose should be stable throughout the study unless it is clinically necessary to adjust the medication.

Exclusion Criteria:

* Dementia not due to probable Alzheimer's disease
* Pregnancy, breastfeeding. The rationale is that retinoids are teratogenic and are excreted in breast milk.
* History of clinically significant stroke
* Modified Hachinski Ischemia score ≥ 4
* Current evidence or history in past two years of epilepsy, seizure, focal brain lesion, head injury with loss of consciousness or DSM IV criteria for any major psychiatric disorder including psychosis, major depression, bipolar disorder, severe alcohol or substance abuse.
* Sensory impairment which would prevent subject from participating in or cooperating with the protocol.
* Use of another investigational agent within two months.
* Evidence of any significant clinical disorder or laboratory finding that renders the participant unsuitable for receiving an investigational new drug including clinically significant or unstable hematologic, hepatic, cardiovascular (including history of ventricular fibrillation or ventricular tachycardia), pulmonary, gastrointestinal, endocrine, metabolic, renal, or other systemic disease or laboratory abnormality. Abnormal liver function test, including AST, ALT, total bilirubin, or prothrombin time. The rationale is that retinoids can be hepatotoxic.
* Participants receiving behavioral medications (including antidepressants, antipsychotics and anxiolytics) must be on stable doses for at least 4 weeks prior to randomization.
* Active neoplastic disease and any medical conditions requiring concurrent immunosuppression.
* Hypertriglyceridemia greater than 500 mg/dL despite statin/fibrate therapy. The rationale is that retinoids can increase lipids, particularly triglyceride and this can lead to pancreatitis.
* Any medical conditions requiring concurrent use of tetracycline, minocycline, or doxycycline. The rationale is due to enhanced risk of increased intracranial pressure.
* Hypersensitivity to retinoids.
* Presence of psychosis or hallucinations at baseline as determined by Neuropsychiatric inventory or Geriatric Depression Scale-short form greater than or equal to five
* Presence of any unstable cardiovascular disease, uncontrolled diabetes, chronic inflammatory or infectious conditions. Retinoids have been associated with chest pain of unclear etiology, increased serum glucose, myelosuppression and increased risk of infection.
* Use of Drugs and supplements such as: Vitamin A supplements beyond 100% RDA, other immunosuppressants (corticosteroids, chemotherapeutic agents, etc.), Warfarin , Fish Oil (DHA)
* Any other disease or medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this clinical trial.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Lerner, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- Parkway Medical Building, Beachwood, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Not anticipated to release subject level data

REFERENCES:
- [Background] Lee HP, Casadesus G, Zhu X, Lee HG, Perry G, Smith MA, Gustaw-Rothenberg K, Lerner A. All-trans retinoic acid as a novel therapeutic strategy for Alzheimer's disease. Expert Rev Neurother. 2009 Nov;9(11):1615-21. doi: 10.1586/ern.09.86. PMID 19903021
- See also: University Hospitals Case Medical Center — http://www.uhhospitals.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from clinical population of PI
Period: Overall Study
Arm/Group | Open Label
Started | 3
Screened | 3 (3 subjects screend and started treatment in open label)
Completed | 0 (Study stopped due to adverse events One subject had transient loss of consciousness - possibly related to treatment One subject declined rapidly and found to have glioblastoma- not rrelated to treatment)
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Open Label
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants] — age>65
  Participants
    <=18 years | 0
    Between 18 and 65 years | 0
    >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 3
impaired cognition due to alzheimer's disease diagnosis [Count of Participants; unit: Participants] | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Six Month Timepoint in the Score on the Alzheimer's Disease Assessment Scale- Cognitive Subscale
Description: Alzheimer's disease Assessment Scale- Cognitive subscale is a scale to measure cognitive function used in dementia clinical trials. No primary outcome data since study was terminated before any participaant completed
Time Frame: 6 months from baseline
Population: Data not collected
Groups:
- Open Label Treatment: All participants will receive Isotretinoin for 24 weeks
Arm/Group | Open Label Treatment
Number analyzed (Participants) | 0

2. Secondary Outcome: Number of Adverse Effects
Description: Any adverse events reported by subject or study partner will be recorded at each visit after screening (Baseline, and visits at week 4, 8, 12, 16, 20, 24, and 28 (four weeks after treatment discontinuation).
Time Frame: 28 weeks
Measure: Number; unit: Number of events
Arm/Group | Open Label
Number analyzed (Participants) | 3
Number of events | 2

ADVERSE EVENTS:
Groups:
- Open Label Treatment: Study terminated due to adverse events leading to PI decision to terminate study
Arm/Group | Open Label Treatment
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 1/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Treatment (N=3)
neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) — Rapid ccognitive decline; found to have glioblastoma
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open Label Treatment (N=3)
loss of consciousness (Nervous system disorders) | 1 (1) — Transient lossw of consciousness in one participant

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes